CLINICAL TRIAL: NCT00386672
Title: Calcium Supplementation for a Healthy Weight- LITE
Brief Title: Calcium Supplementation for a Healthy Weight-Lite (CaSHeW Lite)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Beverage Institute for Health and Wellness (Unknown)
Responsible Party: Principal Investigator, Lee Kaplan MD, PhD, Director, MGH Weight Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-P-000505
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Overweight
Keywords: Calcium; Vitamin D; Weight Loss; Overweight; Obesity; Lite Orange Juice
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lite OJ with Ca and VitD (Experimental): 240ml of reduced energy (lite) OJ beverage fortified with 350mg Ca and 100U VitD, 3 times per day.
  Interventions: Dietary Supplement: Reduced energy (lite) OJ fortified with Calcium and Vitamin D; Behavioral: Nutrition Counseling
- Lite OJ without Ca and VitD (Active Comparator): 240ml of reduced energy (lite) OJ beverage, 3 times per day.
  Interventions: Behavioral: Nutrition Counseling; Dietary Supplement: Reduced energy (lite) OJ without Calcium and Vitamin D

INTERVENTIONS:
Dietary Supplement: Reduced energy (lite) OJ fortified with Calcium and Vitamin D — Three 240ml servings of lite OJ fortified with 350mg Ca and 100U VitD per day.
  Other Names: Minute Maid Light Orange Juice
  Arms: Lite OJ with Ca and VitD
Behavioral: Nutrition Counseling — Individual and group nutritional counseling by a registered dietician.
Dietary Supplement: Reduced energy (lite) OJ without Calcium and Vitamin D — Three 240ml servings of lite OJ without 350mg Ca and 100U VitD per day.
  Other Names: Minute Maid Light Orange Juice
  Arms: Lite OJ without Ca and VitD

SUMMARY:
The purpose of the study is to find out if taking calcium and vitamin D supplements, while following a low-calorie diet, can help people lose weight.

DETAILED DESCRIPTION:
Recent studies suggest that calcium may be important for weight loss, but other studies have not had the same results. The purpose of the study is to find out if taking calcium and vitamin D supplements, while following a low-calorie diet, can help people lose weight.

We will use special orange juice with less calories than regular orange juice. Half of the subjects in this study will drink the study juice (reduced-calorie orange juice) containing extra calcium and vitamin D. The other subjects will drink reduced-calorie orange juice without any extra calcium or vitamin D in it.

Comparisons: We will compare subjects who follow the diet and take calcium and vitamin D supplements to those who only follow the diet.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, between 18 and 65 years of age, who are capable of providing informed consent.
* BMI of 25 to 35 kg/m2.
* Non-smoker (for at least 6 months).
* In good health, as determined by the principal investigator based on medical history and physical examination.
* Clinical laboratory evaluations (including Biochemistry, Hematology, Endocrinology) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator.
* Because of the calorie-restricted diet and radiation exposure from the CT scan, females will be non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile for at least 3 months, or be willing to use an approved method of contraception (which may include use of abstinence; intrauterine device; female condom with spermicide; diaphragm with spermicide; cervical cap with spermicide; oral or transdermal hormonal contraceptives; a condom with spermicide by the sexual partner; or a sterile sexual partner) from 35 days prior to study entry (i.e., Day -1) until 30 days following Study Completion. For all females, the pregnancy test result must be negative at the screening visit and at visits when a CT scan will be done.
* Ability to comprehend and willingness to sign the Informed Consent Form for this study.
* Ability to comply with study restrictions regarding diet and exercise.
* Stable weight (+ 5%) for at least 3 months prior to study entry.

Exclusion Criteria:

* Diabetes mellitus.
* History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders which in the opinion of the investigator would be expected to interfere with the study or increase risk to the subject.
* Participation in any other investigational diet study within 90 days prior to study entry.
* History of a medical or psychological condition or social circumstances that would impair the subject's ability to participate reliably in the study.
* Use within the last six months of medications that can result in significant weight gain or weight loss, including antipsychotics, selective serotonin reuptake inhibitors, anti-epileptic drugs, appetite-suppressants such as phentermine and sibutramine, and the lipase-inhibitor orlistat. (see Appendix 1 for detailed list)
* Active eating disorder.
* History of alcoholism or substance abuse within 5 years prior to study entry.
* Recommendation by a physician to avoid calcium supplements because of a history of kidney stones or other medical condition.
* History of hyperparathyroidism or sarcoidosis.
* Osteoporosis or other medical condition for which a physician has recommended taking a multivitamin or calcium supplementation.
* High calcium intake (more than 2 servings of dairy products per day or taking calcium supplements > 3x/wk ) for 1 month prior to study start date and for duration of study. (If participant is taking calcium supplement > 3x/wk or more than 2 servings of dairy products per day, they are eligible to participate if they agree to stop for 1 month prior to study start date and for the duration of the study. Participants will similarly be asked to stop multivitamins as the majority of these supplements contain calcium.)
* General medical conditions that are well-controlled will not be a basis for exclusion in the study. Subjects with uncontrolled conditions that are not adequately controlled or that might pose an unacceptable risk for participation, as clinically determined by the investigators, will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline and at 16 weeks

SECONDARY OUTCOMES:
Change in visceral adipose tissue mass | Baseline and at 16 weeks
Change in subcutaneous adipose tissue mass | Baseline and at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Kaplan, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Weight Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Wolf AM, Colditz GA. Current estimates of the economic cost of obesity in the United States. Obes Res. 1998 Mar;6(2):97-106. doi: 10.1002/j.1550-8528.1998.tb00322.x. PMID 9545015
- [Background] Davies KM, Heaney RP, Recker RR, Lappe JM, Barger-Lux MJ, Rafferty K, Hinders S. Calcium intake and body weight. J Clin Endocrinol Metab. 2000 Dec;85(12):4635-8. doi: 10.1210/jcem.85.12.7063. PMID 11134120
- [Background] Jacqmain M, Doucet E, Despres JP, Bouchard C, Tremblay A. Calcium intake, body composition, and lipoprotein-lipid concentrations in adults. Am J Clin Nutr. 2003 Jun;77(6):1448-52. doi: 10.1093/ajcn/77.6.1448. PMID 12791622
- [Background] Zemel MB. Regulation of adiposity and obesity risk by dietary calcium: mechanisms and implications. J Am Coll Nutr. 2002 Apr;21(2):146S-151S. doi: 10.1080/07315724.2002.10719212. PMID 11999543
- [Background] Zemel MB, Shi H, Greer B, Dirienzo D, Zemel PC. Regulation of adiposity by dietary calcium. FASEB J. 2000 Jun;14(9):1132-8. PMID 10834935
- [Background] Shi H, Norman AW, Okamura WH, Sen A, Zemel MB. 1alpha,25-Dihydroxyvitamin D3 modulates human adipocyte metabolism via nongenomic action. FASEB J. 2001 Dec;15(14):2751-3. doi: 10.1096/fj.01-0584fje. Epub 2001 Oct 15. PMID 11606486
- [Background] Zemel MB. Role of dietary calcium and dairy products in modulating adiposity. Lipids. 2003 Feb;38(2):139-46. doi: 10.1007/s11745-003-1044-6. PMID 12733746
- [Background] Shi H, Dirienzo D, Zemel MB. Effects of dietary calcium on adipocyte lipid metabolism and body weight regulation in energy-restricted aP2-agouti transgenic mice. FASEB J. 2001 Feb;15(2):291-3. doi: 10.1096/fj.00-0584fje. Epub 2000 Dec 8. PMID 11156940
- [Background] Ye WZ, Reis AF, Dubois-Laforgue D, Bellanne-Chantelot C, Timsit J, Velho G. Vitamin D receptor gene polymorphisms are associated with obesity in type 2 diabetic subjects with early age of onset. Eur J Endocrinol. 2001 Aug;145(2):181-6. doi: 10.1530/eje.0.1450181. PMID 11454514
- [Background] Barger-Lux MJ, Heaney RP, Hayes J, DeLuca HF, Johnson ML, Gong G. Vitamin D receptor gene polymorphism, bone mass, body size, and vitamin D receptor density. Calcif Tissue Int. 1995 Aug;57(2):161-2. doi: 10.1007/BF00298438. PMID 7584878
- [Background] Bell NH, Epstein S, Greene A, Shary J, Oexmann MJ, Shaw S. Evidence for alteration of the vitamin D-endocrine system in obese subjects. J Clin Invest. 1985 Jul;76(1):370-3. doi: 10.1172/JCI111971. PMID 2991340
- [Background] Liel Y, Ulmer E, Shary J, Hollis BW, Bell NH. Low circulating vitamin D in obesity. Calcif Tissue Int. 1988 Oct;43(4):199-201. doi: 10.1007/BF02555135. PMID 3145124
- [Background] Shi H, Norman AW, Okamura WH, Sen A, Zemel MB. 1alpha,25-dihydroxyvitamin D3 inhibits uncoupling protein 2 expression in human adipocytes. FASEB J. 2002 Nov;16(13):1808-10. doi: 10.1096/fj.02-0255fje. Epub 2002 Sep 5. PMID 12223452
- [Background] Sun X, Zemel MB. Role of uncoupling protein 2 (UCP2) expression and 1alpha, 25-dihydroxyvitamin D3 in modulating adipocyte apoptosis. FASEB J. 2004 Sep;18(12):1430-2. doi: 10.1096/fj.04-1971fje. Epub 2004 Jul 1. PMID 15231722
- [Background] Zemel MB, Miller SL. Dietary calcium and dairy modulation of adiposity and obesity risk. Nutr Rev. 2004 Apr;62(4):125-31. doi: 10.1111/j.1753-4887.2004.tb00034.x. PMID 15141427
- [Background] Melanson EL, Sharp TA, Schneider J, Donahoo WT, Grunwald GK, Hill JO. Relation between calcium intake and fat oxidation in adult humans. Int J Obes Relat Metab Disord. 2003 Feb;27(2):196-203. doi: 10.1038/sj.ijo.802202. PMID 12586999
- [Background] Pereira MA, Jacobs DR Jr, Van Horn L, Slattery ML, Kartashov AI, Ludwig DS. Dairy consumption, obesity, and the insulin resistance syndrome in young adults: the CARDIA Study. JAMA. 2002 Apr 24;287(16):2081-9. doi: 10.1001/jama.287.16.2081. PMID 11966382
- [Background] Heaney RP, Davies KM, Barger-Lux MJ. Calcium and weight: clinical studies. J Am Coll Nutr. 2002 Apr;21(2):152S-155S. doi: 10.1080/07315724.2002.10719213. PMID 11999544
- [Background] Rosenblum JL, Castro VM, Moore CE, Kaplan LM. Calcium and vitamin D supplementation is associated with decreased abdominal visceral adipose tissue in overweight and obese adults. Am J Clin Nutr. 2012 Jan;95(1):101-8. doi: 10.3945/ajcn.111.019489. Epub 2011 Dec 14. PMID 22170363